CLINICAL TRIAL: NCT04734522
Title: Assessment of Progressive Lens Designs
Acronym: TBPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Hoya Vision Care (Industry)
Responsible Party: Principal Investigator, Silvia Tavazzi, Professor, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2019-01
Record Dates: First submitted 2021-01-15; First posted 2021-02-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Presbyopia
Keywords: presbyopia; progressive addition lenses
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The specified PAL design wearers (Experimental): Subjects who have been already wearing any from specified design type of PAL
  Interventions: Device: Progressive Additional Lenses (PAL), pre calibrated and made of polymeric material with anti-reflection coating
- The other PAL design wearers (Active Comparator): Subjects who have been already wearing any from the other design type of PAL
  Interventions: Device: Progressive Additional Lenses (PAL), pre calibrated and made of polymeric material with anti-reflection coating

INTERVENTIONS:
Device: Progressive Additional Lenses (PAL), pre calibrated and made of polymeric material with anti-reflection coating — Subjects will be wearing three different PAL designs with different geometries of the optical progression.

SUMMARY:
Non-invasive double-blind randomised comparative study on presbyopic subjects wearing progressive lenses.

DETAILED DESCRIPTION:
Background and rationale:

Nowadays many different types of progressive addition lenses are available for the correction of presbyopia. Progressive addition lenses provide a more natural correction for presbyopic people due to a gradual and progressive increase of lens power from far area through the intermediate portion to the near area. However, some patients still experience adaptation problems.

The primary purpose of the study is to evaluate the preference, adaptability and visual performance of progressive lens designs (up to three designs).

Study procedures:

Each participant is required to wear all pairs of spectacles one after another, each pair for one week.

Each participant will be required to visit the optometry clinic (at University of Milano Bicocca) three times:

Visit #1: Screening based on inclusion criteria, Informed Consent Form (ICF) form signing, Optometric exam and choice of the frame.

Subjects who will pass the inclusion/exclusion screening will be asked to sign the ICF and enrolled for the optometric exam. Subjects will choose the spectacle frame and all individual fitting parameters will be measured for lens' manufacturing.

Visit #2: Subjects will receive three marked pairs of progressive lenses. The three spectacle frames will be adjusted to fit properly on the subject' face. After 10-15 min of wearing of the first pair of lenses, each subject will be asked to answer to a questionnaire.

Visit #3 (last visit): questionnaires should be returned; the last comparison question will be answered during this visit, and subject will choose the best pair.

At the end of the study each participant will be entitled to get one pair of progressive lenses available in the market.

Subject population:

Presbyopic subjects have been already wearing any progressive additional lens (PAL) designs.

Number of Subjects:

40 +/- 2 subjects, the specified PAL design wearers and 40 +/- 2 the other PAL design wearers to be enrolled and signed the informed consent form.

Each subject will be wearing three different PAL designs. Subjects will be asked to choose one pair of spectacles (design) which they like the most.

Randomisation:

This study adopts a stratified permuted block randomisation to reduce an evaluation bias by the wearing sequence and prescriptions. The mean of both eyes' prescriptions is set as a single stratification factor.

Frames:

Each subject will choose a model of spectacle frame. Three identical frames will be taken for each subject.

Lenses:

1. Lenses will be produced in EU
2. Three different lens designs will be tested in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be experienced progressive lens designs wearers who have worn their current prescription for at least the last one month.
2. PAL wearers with 14 mm corridor
3. Age: 45 to 70 years old
4. Best Corrected Monocular visual Acuity (decimal) both at distance and near ≥ 1.0;
5. Normal binocular vision at distance & near:

   * no strabismus on cover test,
   * no fixation disparity (Mallett aligning prism of less than 2Δ horizontally or vertically) at near
   * stereoacuity of 60" or better at near;
6. New prescription (found at visit #1) is in the range:

   * Spherical power: up to +/-6.00;
   * Cylindrical power: minus cylinder ≤ 2.5D;
   * Addition: 1.50-2.50D;
   * Difference in the power (spherical equivalent) between eyes: up to 2.0D
7. Understanding and speaking Italian or English to be able to answer questionnaires
8. Giving a written consent to participate in the study

Exclusion Criteria:

1. First prescription for progressive lenses.
2. Prescription found during visit#1 varies from current prescription more than 0.50D in any meridian
3. Wearing Single Vision lenses with accommodative support
4. Double vision or prismatic prescription in current glasses;
5. Known ocular disease including strabismus, any pathology, any eye surgeries that may affect visual acuity
6. Use of systemic or ocular medications that are likely to affect vision
7. Balance problem/vertigo problem
8. Concurrent participation in other vision-related research

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the preference among progressive lens designs | Entire study duration (approx. 4 weeks)
  Evaluate the preference among progressive lens designs through a "First impression questionnaire" after 10-15 minutes of wearing each of the 3 PALs, a "Final satisfaction questionnaire" after 1 week of use of each of the 3 PALs and a "Comparison questionnaire" at the end of the three trial periods of all the three types of PALs.

SECONDARY OUTCOMES:
Evaluate the adaptability of progressive lens designs. | Entire study duration (approx. 4 weeks)
  Evaluate adaptability of progressive lens designs through a "Final satisfation questionnaire" after one week of use of each of the three PALs.
Evaluate visual performance of progressive lens designs. | Entire study duration (approx. 4 weeks)
  Evaluate the visual performance of progressive lens designs measured both after 10-15 minutes of wear and after one week by psychophysical analysis (visual acuity at high contrast at near and at distance, rate/accuracy of reading test at high contrast and at near).

CONTACTS AND LOCATIONS:
Locations (1):
- Optics and Optometry of Milano-Bicocca (COMiB), Department of Materials Science - University of Milano-Bicocca, Milan, Italy